CLINICAL TRIAL: NCT00005980
Title: A Randomized Phase II Study of Two Different Schedules of Caelyx in Metastatic Breast Cancer
Brief Title: Comparison of Two Regimens of Liposomal Doxorubicin in Treating Women With Metastatic Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Responsible Party: Sponsor
Allocation: Randomized | Purpose: Treatment
Other Study IDs: EORTC-10993-16998; EORTC-IDBBC-10993; ECSG-10993; PAMM-10993
Record Dates: First submitted 2000-07-05; First posted 2003-01-27 (Estimated); Last update posted 2012-07-18 (Estimated); Status verified 2012-07

CONDITIONS: Breast Cancer
Keywords: stage IV breast cancer; recurrent breast cancer
MeSH Terms: conditions — Breast Neoplasms

INTERVENTIONS:
Drug: pegylated liposomal doxorubicin hydrochloride

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. It is not yet known which regimen of liposomal doxorubicin is more effective for metastatic breast cancer.

PURPOSE: Randomized phase II trial to compare the effectiveness of two regimens of liposomal doxorubicin in treating women who have metastatic breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the response rate in women with metastatic breast cancer treated with two different dose schedules of doxorubicin HCL liposome.
* Assess the side effects of these treatment regimens in this patient population.
* Determine the duration of response in these patients treated with these regimens.
* Assess the concentration of doxorubicin in tumor tissue in patients with easily accessible metastases.

OUTLINE: This is a randomized, multicenter study. Patients are stratified according to participating center, performance status (0-1 vs 2), visceral disease (yes vs no), available lesions for biopsy (yes vs no), prior adjuvant anthracyclines (yes vs no), and prior chemotherapy for advanced disease (yes vs no). Patients are randomized to one of two treatment arms.

* Arm I: Patients receive doxorubicin HCL liposome IV over 1 hour every 6 weeks.
* Arm II: Patients receive doxorubicin HCL liposome IV over 1 hour every 4 weeks. Treatment continues for at least 36 weeks in the absence of disease progression or unacceptable toxicity.

Patients are followed every 3 months.

PROJECTED ACCRUAL: A total of 64-100 patients (32-50 per treatment arm) will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically proven progressive or recurrent metastatic breast cancer
* Bidimensionally measurable disease with at least one target lesion

  * If previously irradiated lesions:

    * No preirradiated only lesions
    * Clear progression prior to study
    * New lesions in a previously irradiated region allowed
* Refusal of or medical contraindication to standard anthracycline containing regimen
* Hormone receptor status:

  * Not specified

PATIENT CHARACTERISTICS:

Age:

* Any age

Sex:

* Female

Menopausal status:

* Not specified

Performance status:

* ECOG 0-2

Life expectancy:

* Not specified

Hematopoietic:

* Neutrophil count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3

Hepatic:

* Bilirubin normal
* Transaminases less than 2 times upper limit of normal

Renal:

* Creatinine normal

Cardiovascular:

* Left ventricular ejection fraction normal by echocardiography or MUGA scan
* No significant cardiac history including:

  * Clinically significant atrial or ventricular arrhythmias requiring treatment
  * Medically controlled congestive heart failure
  * Significant angina or clinically and/or electrocardiographically documented myocardial infarction within the past year
  * Clinically significant valvular disease

Other:

* No other prior or concurrent malignancy within the past 5 years except contralateral breast cancer, or adequately treated basal cell skin cancer or carcinoma in situ of the cervix
* No psychological, familial, sociological, or geographical condition that would preclude study
* Not pregnant or nursing
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* See Disease Characteristics
* Prior adjuvant chemotherapy allowed if total doxorubicin dose is no greater than 300 mg/m2, total epirubicin dose is no greater than 450 mg/m^2, and total mitoxantrone dose is no greater than 75 mg/m^2
* No greater than one regimen of prior chemotherapy for metastatic disease
* No prior anthracyclines for metastatic disease
* No other concurrent cytotoxic therapy

Endocrine therapy:

* No concurrent hormonal therapy
* At least 4 weeks since prior progestins, estrogens, or androgens

Radiotherapy:

* See Disease Characteristics
* Concurrent palliative radiotherapy allowed if sole target lesion is outside irradiated field

Surgery:

* Not specified

Other:

* Concurrent bisphosphonates for metastatic bone disease and hypercalcemia secondary to malignancy allowed if bony lesions not only target lesion
* No other concurrent investigational therapy

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 116 (Actual)
Dates: Start 2000-04; Primary Completion 2002-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert E. Coleman, MD, FRCP, Study Chair — Cancer Research Centre at Weston Park Hospital; Maurizio D'Incalci, MD, Study Chair — Mario Negri Institute for Pharmacological Research; Christian Dittrich, MD, Study Chair — Ludwig Boltzmann Institute for Applied Cancer Research at Kaiser Franz Josef Hospital
Locations (14):
- Ludwig Boltzmann - Institute for Applied Cancer Research, Vienna, Austria
- France (4):
  - Institut Bergonie, Bordeaux
  - Centre Jean Perrin, Clermont-Ferrand
  - Institut Curie - Section Medicale, Paris
  - Centre Henri Becquerel, Rouen
- University of Ioannina, Ioannina, Greece
- Rabin Medical Center - Beilinson Campus, Petah Tikva, Israel
- Italy (2):
  - Mario Negri Institute for Pharmacological Research, Milano (Milan)
  - Istituti Fisioterapici Ospitalieri - Roma, Rome
- Netherlands (2):
  - Academisch Ziekenhuis Groningen, Groningen
  - University Medical Center Nijmegen, Nijmegen
- Hospital Universitario 12 de Octubre, Madrid, Spain
- Clinique De Genolier, Genolier, Switzerland
- Royal Marsden NHS Trust, London, England, United Kingdom

REFERENCES:
- [Background] Biganzoli L, Coleman R, Minisini A, Hamilton A, Aapro M, Therasse P, Mottino G, Bogaerts J, Piccart M. A joined analysis of two European Organization for the Research and Treatment of Cancer (EORTC) studies to evaluate the role of pegylated liposomal doxorubicin (Caelyx) in the treatment of elderly patients with metastatic breast cancer. Crit Rev Oncol Hematol. 2007 Jan;61(1):84-9. doi: 10.1016/j.critrevonc.2006.07.008. Epub 2006 Nov 20. PMID 17116400
- [Result] Coleman RE, Biganzoli L, Canney P, Dirix L, Mauriac L, Chollet P, Batter V, Ngalula-Kabanga E, Dittrich C, Piccart M. A randomised phase II study of two different schedules of pegylated liposomal doxorubicin in metastatic breast cancer (EORTC-10993). Eur J Cancer. 2006 May;42(7):882-7. doi: 10.1016/j.ejca.2005.12.011. Epub 2006 Mar 7. PMID 16520033